CLINICAL TRIAL: NCT03287622
Title: Scenario-tailored Opioid Messaging Program (STOMP): An Interactive Intervention to Prevent Opioid-related Adverse Drug Events in Children and Adolescents
Brief Title: Evaluation of an Interactive Opioid Risk Education Program (STOMP) for Parents
Acronym: STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Terri Voepel-Lewis, Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 00127009; 1R01DA044245-01A1 (NIH)
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative; Medication Adherence; Opioid Use; Knowledge, Attitudes, Practice; Risk Reduction Behavior
MeSH Terms: conditions — Pain, Postoperative; Medication Adherence; Behavior; Risk Reduction Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Four-armed, randomized, control, factorial design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Group assignment will be coded for parents and data collectors. Parents will be blinded to whether the information they receive is the Intervention vs. Control.
  Group assignment will coded on data entry and unblinded after analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Education Intervention + Nudge (Experimental): This group will receive BOTH the scenario-tailored STOMP educational feedback AND the behavioral Nudge intervention
  Interventions: Behavioral: Educational Intervention; Behavioral: Nudge
- Standard of Care + Nudge (Experimental): This group will receive routine, standard of care information AND the behavioral Nudge intervention
  Interventions: Behavioral: Nudge
- Educational Intervention no Nudge (Experimental): This group will receive scenario-tailored opioid message (STOMP) feedback and NO behavioral nudge intervention.
  Interventions: Behavioral: Educational Intervention
- Standard of Care no Nudge (No Intervention): This group will receive only standard of care information and NO behavioral nudge intervention.

INTERVENTIONS:
Behavioral: Educational Intervention — This intervention provides scenario-tailored opioid risk message feedback immediately following interactive analgesic decision-making exercises.
  Other Names: STOMP Intervention
  Arms: Education Intervention + Nudge; Educational Intervention no Nudge
Behavioral: Nudge — Behavioral Nudge in this study is a simple, take-home kit (ziplock baggy of used coffee grounds) to be used to dispose of left-over prescription opioids
  Arms: Education Intervention + Nudge; Standard of Care + Nudge

SUMMARY:
Millions of children and adolescents are prescribed opioid pain relievers each year, placing them at risk for serious adverse events and misuse in the home setting. Parents who manage these medicines, therefore, need to recognize opioid-related risks and make decisions that will both reduce these risks yet ensure effective pain relief for their children. The proposed research will evaluate new strategies to help parents learn about opioid risks, make safe and effective analgesic decisions, and develop and demonstrate safe drug management behaviors. 840 parents and their children who are undergoing an elective surgical procedure will be recruited. Parents will be randomized to receive the new educational and practical behavioral strategy or routine information. Parents' knowledge and perceptions will be evaluated at baseline and at critical times after surgery. Parents' opioid handling and administration will also be assessed.

DETAILED DESCRIPTION:
The overarching goal of this research is to improve opioid analgesic safety and efficacy by optimizing opioid risk recognition, informed analgesic decision-making, and drug storage/disposal behaviors among parents of youth who are prescribed these agents for home use. The study aims are to determine whether the Scenario-Tailored Opioid Messaging Program (STOMP) will: 1) Improve parents' opioid risk understanding and their analgesic decision-making; 2) Enhance parents' analgesic self-efficacy, analgesic use, storage behaviors and their children's pain outcomes, and 3) To demonstrate that the STOMP plus provision of a simple method to get rid of left-over opioids will effectively nudge parents to safely dispose of left-over opioid analgesics. Parents whose children are prescribed opioids for acute, short-lived pain after surgery will be randomly assigned to receive our interventions or a routine provider informational interaction at the time of opioid prescribing. Parents will be surveyed about their opioid familiarity, knowledge, risk perceptions and common analgesic decision-making at baseline and after hospital discharge. Parents will also record their child's pain medication use and symptoms after discharge. Data will be analyzed to determine whether the STOMP educational intervention with or without the behavioral nudge intervention will enhance parents' risk perceptions, their decision-making skills and their opioid handling behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parent (>=21yr) and child (5-17 yr) (dyad) who lives in the home and is prescribed an opioid for postoperative pain management
* English speaking

Exclusion Criteria:

* Child is undergoing a non-elective procedure
* Child cannot self-report pain levels (i.e., is cognitively impaired)
* Child has a hematologic/oncologic condition
* Child has a kidney or liver conditions that precludes the usual analgesic prescription pattern (opioid plus a non-opioid)
* Child has been taking opioids for prolonged pain pre-operatively (>2 weeks)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Voepel-Lewis, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voepel-Lewis T, Boyd CJ, Tait AR, McCabe SE, Zikmund-Fisher BJ. A Risk Education Program Decreases Leftover Prescription Opioid Retention: An RCT. Am J Prev Med. 2022 Oct;63(4):564-573. doi: 10.1016/j.amepre.2022.04.035. Epub 2022 Jul 28. PMID 35909029
- [Derived] Voepel-Lewis T, Farley FA, Grant J, Tait AR, Boyd CJ, McCabe SE, Weber M, Harbagh CM, Zikmund-Fisher BJ. Behavioral Intervention and Disposal of Leftover Opioids: A Randomized Trial. Pediatrics. 2020 Jan;145(1):e20191431. doi: 10.1542/peds.2019-1431. PMID 31871245

RESULTS

PARTICIPANT FLOW:
Groups:
- Education Intervention: This group will receive the scenario-tailored STOMP educational feedback.
  Educational Intervention: This intervention provides scenario-tailored opioid risk message feedback immediately following interactive analgesic decision-making exercises.
- Standard of Care: This group will receive routine, standard of care information
Period: Overall Study
Arm/Group | Education Intervention | Standard of Care
Started | 356 | 356
Sub-randomized to Nudge/NoNudge | 253 | 266
Completed | 298 | 308
Not Completed | 58 | 48
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 27 | 15
Not completed — No prescripion after surgery | 28 | 31
Not completed — prolonged Length of stay | 2 | 0
Not completed — surgery related | 0 | 2

BASELINE CHARACTERISTICS:
Population: 298 subjects (84%) completed surveys required for analysis in the INTERVENTION GROUP.
  308 subjects (87%) completed surveys required for analysis in the STANDARD OF CARE GROUP
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Intervention | Standard of Care | Total
Number analyzed (Participants) | 298 | 308 | 606
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 298 | 308 | 606
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 298 subjects completed surveys required for analysis in the INTERVENTION GROUP. 308 subjects completed surveys required for analysis in the STANDARD OF CARE GROUP
  Participants
    Female | 252 | 241 | 493
    Male | 46 | 67 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 298 subjects completed surveys required for analysis in the INTERVENTION GROUP. 308 subjects completed surveys required for analysis in the STANDARD OF CARE GROUP
  Participants
    Hispanic or Latino | 9 | 10 | 19
    Not Hispanic or Latino | 289 | 298 | 587
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 298 subjects completed surveys required for analysis in the INTERVENTION GROUP. 308 subjects completed surveys required for analysis in the STANDARD OF CARE GROUP
  Participants
    American Indian or Alaska Native | 2 | 3 | 5
    Asian | 7 | 6 | 13
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 19 | 18 | 37
    White | 262 | 267 | 529
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 7 | 14 | 21
Education Level [Count of Participants; unit: Participants]
  Some HS or HS complete | 38 | 31 | 69
  Some College | 60 | 57 | 117
  Assoc. Degree or Trade School | 62 | 54 | 116
  4 Year College Graduate | 76 | 84 | 160
  Graduate School | 62 | 82 | 144

OUTCOME MEASURES:

1. Primary Outcome: Opioid-related Risk Knowledge
Description: Number of parent participants who became aware (binary) of serious opioid-related adverse effect (over sedation)
Time Frame: Day 3 follow-up assessment
Population: These parents completed at least one follow-up assessment for risk awareness
Measure: Count of Participants; unit: Participants
Groups:
- Education Intervention: This group received the scenario-tailored STOMP educational feedback.
  Educational Intervention: This intervention provides scenario-tailored opioid risk message feedback immediately following interactive analgesic decision-making exercises.
- Standard of Care Education: This group received routine, standard of care information.
Arm/Group | Education Intervention | Standard of Care Education
Number analyzed (Participants) | 296 | 308
Participants | 287 | 289

2. Primary Outcome: Opioid Risk Perception
Description: Change in parent's perceived risk of keeping/sharing opioids (misuse) (Risk perceptions measured on scale from -4 to +4 where higher number reflects higher perception of riskiness; the outcome is measured as change in risk perception - positive change indicates that risk perception became greater)
Time Frame: Mean difference in score from baseline to follow-up assessments (Days 3 & 14)
Population: 296 in the Interventional Group completed at least one follow-up assessment and 281 in the Standard of Care group did so.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Standard of Care: This group received routine, standard of care information
Arm/Group | Education Intervention | Standard of Care
Number analyzed (Participants) | 296 | 281
units on a scale
  Mean difference in perceived riskiness of keeping/sharing opioids day 3 | 0.35 [0.07 to 0.63] | 0.12 [-0.06 to 0.29]
  Change in perceived riskiness keeping/sharing day 14 | 0.28 [0.07 to 0.50] | 0.14 [-0.06 to 0.33]

3. Secondary Outcome: Opioid Disposal Behavior
Description: Number of parents (and percentage) who disposed of left-over opioids after use
Time Frame: Day 14 (or after course completion)
Population: This subgroup analysis included parents that were randomized to four groups.
Measure: Count of Participants; unit: Participants
Groups:
- Nudge + Educational Intervention: This group received BOTH the scenario-tailored STOMP educational feedback AND the behavioral Nudge intervention
  Nudge: Behavioral Nudge in this study is a simple, take-home kit (ziplock baggy of used coffee grounds) to be used to dispose of left-over prescription opioids
- Nudge + Standard of Care: This group received routine, standard of care information AND the behavioral Nudge intervention
  Nudge: Behavioral Nudge in this study is a simple, take-home kit (ziplock baggy of used coffee grounds) to be used to dispose of left-over prescription opioids
- Educational Intervention Only (No Nudge): This group received scenario-tailored opioid message (STOMP) feedback and NO behavioral nudge intervention.
  Educational Intervention: This intervention provides scenario-tailored opioid risk message feedback immediately following interactive analgesic decision-making exercises.
- Standard of Care Only (No Nudge): This group received only standard of care information and NO behavioral nudge intervention.
Arm/Group | Nudge + Educational Intervention | Nudge + Standard of Care | Educational Intervention Only (No Nudge) | Standard of Care Only (No Nudge)
Number analyzed (Participants) | 124 | 131 | 129 | 133
Participants | 48 | 44 | 40 | 25

4. Secondary Outcome: Pain Interference (PROMIS)
Description: The Parents PROMIS Pain Interference measure was used to capture pain interference with functioning (score range 0-30 with higher number indicating worse pain interference)
Time Frame: Day 14
Population: These are the parents that recorded a value in the follow-up diary/survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Standard of Care
Number analyzed (Participants) | 271 | 292
units on a scale | 8.63 (8.39) | 8.06 (8.06)

5. Secondary Outcome: Analgesic Self-Efficacy
Description: Survey measures how confident the parent is in managing pain and opioid-related adverse events (score range 0-35; higher = more efficacy)
Time Frame: Efficacy scores Day 14
Population: Completion of at least one follow-up efficacy assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Standard of Care
Number analyzed (Participants) | 298 | 308
units on a scale | 32.5 (3.22) | 32.2 (3.25)

6. Secondary Outcome: Analgesic Use / Adherence
Description: Total number of opioid doses administered
Time Frame: Day 14
Population: These parents completed follow-up data regarding doses administered at home (completed diary or survey)
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Education Intervention | Standard of Care
Number analyzed (Participants) | 292 | 271
Doses | 8.6 (10.3) | 7.9 (8.6)

7. Secondary Outcome: Analgesic Decision Competency
Description: Number of participants who made the scenario-based decision to administer opioid to excessively sedated child
Time Frame: Day 3
Population: Parents who completed at scenario decisions in Day 3 follow-up survey
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care Only: This group received routine, standard of care information
Arm/Group | Education Intervention | Standard of Care Only
Number analyzed (Participants) | 298 | 308
Participants | 43 | 64

ADVERSE EVENTS:
Time Frame: All adverse events within 30 days of enrollment were recorded.
Description: All adverse effects were recorded according to the definition from clinicaltrials.gov. Of particular interest for this study were all analgesic-related side effects and parent calls and any return to the hospital. Clinic notes (30 days) were reviewed for surgical and analgesic-related calls or return visits to the clinic or hospital.
Arm/Group | Education Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/308
Serious Adverse Events (participants affected / at risk) | 4/298 | 3/308
Other Adverse Events (participants affected / at risk) | 0/298 | 0/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Education Intervention (N=298) | Standard of Care (N=308)
Dehydration (Metabolism and nutrition disorders) | 1 (298) | 1 (308) — dehydration due to poor fluid intake at home
Postoperative hemorrhage (Surgical and medical procedures) | 1 (298) | 1 (308) — Bleeding due to otorhinolaryngology procedure (postoperative bleeding)
Suspected postoperative infection (Surgical and medical procedures) | 0 (0) | 1 (308) — Fever, elevated white blood cell count; treated for postoperative infection
Deep vein thrombosis (Blood and lymphatic system disorders) | 1 (298) | 0 (0) — deep vein thrombosis after ortho surgery; treated with anticoagulation therapy
Adverse Drug Reaction (General disorders) | 1 (298) | 0 (0) — Child had reaction to a medication used for underlying condition (present preoperatively)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03287622/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03287622/Prot_SAP_001.pdf